CLINICAL TRIAL: NCT01870505
Title: A Phase I Trial of BYL719 Plus Letrozole or Exemestane for Patients With Hormone-Receptor Positive Locally-Advanced Unresectable or Metastatic Breast Cancer
Brief Title: BYL719 Plus Letrozole or Exemestane for Patients With Hormone-Receptor Positive Locally-Advanced Unresectable or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-027
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2022-03

CONDITIONS: Metastatic or Locally-advanced Unresectable Breast Cancer
Keywords: BYL719; Letrozole; Exemestane; 13-027
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Alpelisib; Letrozole; exemestane

ARMS (4):
- Arm A: BYL719 plus Letrozole (Experimental): For both the dose-finding phase and the expansion phase, patients may have stable or progressive disease on letrozole, and BYL719 will be added. A treatment cycle will consist of 28 days. Treatment doses for each AI will be fixed at the established dose. Patients will continue on treatment until progression of disease or unacceptable toxicity. The initial scan interval to assess disease status will be every two cycles (8 weeks) for the first four cycles (16 weeks), and then every 3rd cycle (12 weeks) thereafter.
  Interventions: Drug: BYL719; Drug: Letrozole
- Arm B: BYL719 plus Exemestane (Experimental): For both the dose-finding phase and the expansion phase, patients may have stable or progressive disease on Exemestane, and BYL719 will be added. A treatment cycle will consist of 28 days. Treatment doses for each AI will be fixed at the established dose. Patients will continue on treatment until progression of disease or unacceptable toxicity. The initial scan interval to assess disease status will be every two cycles (8 weeks) for the first four cycles (16 weeks), and then every 3rd cycle (12 weeks) thereafter.
  Interventions: Drug: BYL719; Drug: Exemestane
- Arm C: BYL719 plus Letrozole (Experimental): For both the dose-finding and expansion phases of Arms C and D, patients may have stable or progressive disease on letrozole or exemestane, and BYL719 will be added.Letrozole 2.5mg orally once daily with BYL719 given on days 1-7 and 15-21 of a 28 day cycle. The starting dose of BYL719 in Arms C will be 250mg daily. Patients who are on study under Amendment 13, the scan interval will become every 4th cycle (16 weeks ±4 weeks) from their last scan.
  Interventions: Drug: BYL719; Drug: Letrozole
- Arm D: BYL719 plus Exemestane (Experimental): For both the dose-finding and expansion phases of Arms C and D, patients may have stable or progressive disease on letrozole or exemestane, and BYL719 will be added. Exemestane 25mg orally once daily BYL719 Days 1-5, 8-12, 15-19, 22-26 of 28 day cycle. For Arm D, the established dose is 350mg for BYL719, 10 patients will be assigned to the corresponding arm in the expansion phase of the study. Patients who are on study under Amendment 13, the scan interval will become every 4th cycle (16 weeks ±4 weeks) from their last scan.
  Interventions: Drug: BYL719; Drug: Exemestane

INTERVENTIONS:
Drug: BYL719
Drug: Letrozole
  Arms: Arm A: BYL719 plus Letrozole; Arm C: BYL719 plus Letrozole
Drug: Exemestane
  Arms: Arm B: BYL719 plus Exemestane; Arm D: BYL719 plus Exemestane

SUMMARY:
The purpose of this study is to test the safety of a drug called BYL719 at different dose levels. The investigators want to find out what effects, good and/or bad, BYL719 has on the patient and breast cancer. BYL719 will be given with either letrozole or exemestane to patients with HR+ locally-advanced or metastatic breast cancer. When the recommended phase II dose of BYL719 in combination with letrozole or exemestane has been determined in the dose-finding phase, an additional 10 patients will be enrolled onto each arm in an expansion phase of the study. The purpose of the expansion phase is to further define the safety and feasibility of BYL719 in combination with letrozole or exemestane at the recommended phase II dose, and to estimate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18 years
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Willing and able to consent for biopsy of locally-advanced or metastatic breast cancer prior to treatment
* Metastatic or locally-advanced unresectable breast cancer (includes metastatic or locally-advanced unresectable breast cancer which is diagnosed while on adjuvant letrozole or exemestane)
* Histologically documented HR+ breast cancer in either the primary or metastatic setting, as defined by ER or PR ≥ 1%; results from the local lab are acceptable. Eligibility will not be affected by HER2 status.
* The most recent treatment prior to enrollment must be one of the following (duration of treatment ≥2 weeks), and must have been adequately tolerated according the treating physician's judgment:
* Letrozole
* Exemestane
* Exemestane + everolimus (everolimus must be discontinued for ≥ 3 weeks prior to starting study treatment)
* Letrozole or exemestane in combination with an experimental agent(s) on a clinical trial, provided that the experimental agent(s) is not a PI3K inhibitor or AKT inhibitor (experimental agent(s) must be discontinued for ≥ 3 weeks prior to starting study treatment)
* Any number of prior endocrine therapies (including tamoxifen, fulvestrant and/or aromatase inhibitors in either the adjuvant or metastatic setting) and any number of prior chemotherapy regimens. Anti-cancer systemic therapy, such as chemotherapy or biologics or endocrine therapy, other than the AI, must be discontinued for ≥ 3 weeks prior to starting study treatment.
* For the dose-finding phase, patients must also have stable disease OR progression of disease on the most recent treatment. For the expansion phase, patients must have progression of disease on the most recent treatment. Progression of disease is defined as new or worsening disease on objective imaging. Progression of disease includes recurrence diagnosed while on adjuvant letrozole or exemestane.
* Postmenopausal women, as defined by one of the following (estradiol assay cutoff takes into account that the patient is on aromatase inhibitor therapy):
* Age ≥ 55 years and one year or more of amenorrhea
* Age < 55 years and one year or more of amenorrhea, with an estradiol assay within the post-menopausal range
* Age < 55 years with prior hysterectomy but intact ovaries, with an estradiol assay within the post-menopausal range
* Surgical menopause with bilateral oophorectomy
* Ovarian suppression with a LH-RH agonist, with an estradiol assay within the post-menopausal range at baseline and periodically on-study Measurable or non-measurable disease per RECIST criteria v1.1
* ECOG performance status 0-1
* Adequate organ function, as defined by all of the following:

Hematologic parameters:

* Absolute neutrophil count (ANC) ≥ 1500/μl (without growth factor support)
* Platelets ≥ 100,000/μl (no transfusion allowed within 2 weeks)
* Hemoglobin ≥ 9.0 g/dl (may be reached by transfusion)
* Liver function:
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) unless attributable to Gilbert's syndrome
* AST ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present
* ALT ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present

Kidney function:

* Creatinine ≤ 1.5 ULN
* Endocrine function:
* Fasting plasma glucose <140 mg/dl (may be on antiglycemic agents other than insulin). Fasting glucose measurement must be obtained at least 8 hours after the most recent caloric intake.
* Ability to swallow oral medication
* Willing to discontinue all herbal preparations / medications at least 7 days prior to the first dose of study drug and throughout the study. These include, but not limited to,St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.

Exclusion Criteria:

* Pregnant patients or women who are breast-feeding (patients must be postmenopausal, see Section 6.1.9)

Patients with central nervous system (CNS) involvement may participate if:

* Clinically stable with respect to the CNS tumor at the time of screening and >4 weeks from prior therapy completion (including radiation and/or surgery) to the start of study treatment
* Not receiving steroid therapy
* Not receiving enzyme inducing anti-epileptic medications that were started for brain metastases (these include carbamazepine, phenytoin, phenobarbital, primidone, oxcarbazepine, topiramate, and vigabatrin) Prior PI3K inhibitor or AKT inhibitor (patients previously treated with everolimus are eligible, see rationale in Section 3.6)
* History of toxicity to the most recent AI (letrozole or exemestane) that warrants cessation of the AI
* Patients who have received radiotherapy ≤ 2 weeks prior to starting study treatment
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study treatment, who have not recovered from side effects of such procedure
* Uncontrolled diabetes (as defined by fasting glucose ≥ 140mg/dL) and/or insulin-dependent diabetes. Fasting glucose measurement must be obtained at least 8 hours after the most recent caloric intake. Patients currently requiring the use of antiglycemic agents (other than insulin) may be enrolled if fasting glucose <140mg/dL.
* Current need for chronic corticosteroid therapy (≥10mg of prednisone daily or an equivalent dose of other corticosteroid), or patients who have received systemic corticosteroids ≤ 2 weeks prior to starting study drug
* Current therapeutic anticoagulation with warfarin (or coumarin derivatives) Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment
* Clinically significant cardiac disease or impaired cardiac function, such as:
* Congestive heart failure requiring treatment (e.g., New York Heart Association Class II, III or IV) Acute coronary syndromes < 3 months prior to screening (including myocardial infarction, unstable angina, coronary artery bypass graft, coronary angioplasty, or stenting)
* Uncontrolled arterial hypertension defined by blood pressure > 140/100 mm Hg at rest (average of 3 consecutive readings)
* History or current evidence of unstable, clinically significant cardiac arrhythmias or patients that require medications with a narrow therapeutic window, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high-Grade/complete AV-blockage
* Corrected QT interval (QTc) > 480 msec on screening ECG Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment (see Section 9.6.3 and Appendix F)
* Impaired gastrointestinal function or poorly controlled gastrointestinal disease that may significantly alter the absorption of oral BYL719 (e.g. Crohn's disease, ulcerative colitis, malabsorption syndrome, small bowel resection, uncontrolled nausea or vomiting, or grade ≥ 3 diarrhea of any etiology) based on treating physician assessment
* Patients may not have a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarat Chandarlapaty, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Razavi P, Dickler MN, Shah PD, Toy W, Brown DN, Won HH, Li BT, Shen R, Vasan N, Modi S, Jhaveri K, Caravella BA, Patil S, Selenica P, Zamora S, Cowan AM, Comen E, Singh A, Covey A, Berger MF, Hudis CA, Norton L, Nagy RJ, Odegaard JI, Lanman RB, Solit DB, Robson ME, Lacouture ME, Brogi E, Reis-Filho JS, Moynahan ME, Scaltriti M, Chandarlapaty S. Alterations in PTEN and ESR1 promote clinical resistance to alpelisib plus aromatase inhibitors. Nat Cancer. 2020 Apr;1(4):382-393. doi: 10.1038/s43018-020-0047-1. Epub 2020 Mar 23. PMID 32864625
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- DOSE FINDING PHASE, Arm A, Cohort 0: DOSE FINDING PHASE, Arm A, Cohort 0: BYL719 300mg PO, Letrozole 2.5mg PO
- DOSE FINDING PHASE, Arm A, Cohort -1: DOSE FINDING PHASE, Arm A, Cohort -1: BYL719 250 mg PO, Letrozole 2.5mg PO
- DOSE FINDING PHASE, Arm B, Cohort 0: DOSE FINDING PHASE, Arm B, Cohort 0: BYL719 300mg PO, Exemestane 25mg PO
- Arm D: Arm D : Exemestane 25 mg PO + BYL719 MTD: 350mg PO
- Dose Finding Phase, Arm C, Cohort 0: Dose Finding Phase, Arm C, Cohort 0: Letrozole 2.5mg PO daily & BYL719 250 mg 7days on and 7days off.
- Dose Finding Phase, Arm C, Cohort 1: Dose Finding Phase, Arm C, Cohort 1: Letrozole 2.5mg PO daily & BYL719 300 mg 7days on and 7days off.
- Dose Finding Phase, Arm D, Cohort 0: Dose Finding Phase, Arm D, Cohort 0: Exemestane 25mg PO daily & BYL719 250 mg 5days on and 2days off.
- Dose Finding Phase, Arm D, Cohort 1: Dose Finding Phase, Arm D, Cohort 1: Exemestane 25mg PO daily & BYL719 300 mg 5days on and 2days off.
- Dose Finding Phase, Arm D, Cohort 2: Dose Finding Phase, Arm D, Cohort 2: Exemestane 25mg PO daily & BYL719 350 mg 5days on and 2days off.
Period: Overall Study
Arm/Group | DOSE FINDING PHASE, Arm A, Cohort 0 | DOSE FINDING PHASE, Arm A, Cohort -1 | DOSE FINDING PHASE, Arm B, Cohort 0 | Arm D | Dose Finding Phase, Arm C, Cohort 0 | Dose Finding Phase, Arm C, Cohort 1 | Dose Finding Phase, Arm D, Cohort 0 | Dose Finding Phase, Arm D, Cohort 1 | Dose Finding Phase, Arm D, Cohort 2
Started | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7
Completed | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DOSE FINDING PHASE, Arm A, Cohort 0: Period 1: DOSE FINDING PHASE, Arm A, Cohort 0: BYL719 300mg PO, Letrozole 2.5mg PO
- DOSE FINDING PHASE, Arm A, Cohort -1: Period 2: DOSE FINDING PHASE, Arm A, Cohort -1: BYL719 250 mg PO, Letrozole 2.5mg PO
- DOSE FINDING PHASE, Arm B, Cohort 0: Period 1: DOSE FINDING PHASE, Arm B, Cohort 0: BYL719 300mg PO, Exemestane 25mg PO
- Dose Finding Phase, Arm C, Cohort 0: Period 1: Dose Finding Phase, Arm C, Cohort 0: Letrozole 2.5mg PO daily & BYL719 250 mg 7days on and 7days off.
- Dose Finding Phase, Arm C, Cohort 1: Period 2: Dose Finding Phase, Arm C, Cohort 1: Letrozole 2.5mg PO daily & BYL719 300 mg 7days on and 7days off.
- Dose Finding Phase, Arm D, Cohort 0: Period 1: Dose Finding Phase, Arm D, Cohort 0: Exemestane 25mg PO daily & BYL719 250 mg 5days on and 2days off.
- Dose Finding Phase, Arm D, Cohort 1: Period 2: Dose Finding Phase, Arm D, Cohort 1: Exemestane 25mg PO daily & BYL719 300 mg 5days on and 2days off.
- Dose Finding Phase, Arm D, Cohort 2: Period 3: Dose Finding Phase, Arm D, Cohort 2: Exemestane 25mg PO daily & BYL719 350 mg 5days on and 2days off.
- Total: Total of all reporting groups
Arm/Group | DOSE FINDING PHASE, Arm A, Cohort 0 | DOSE FINDING PHASE, Arm A, Cohort -1 | DOSE FINDING PHASE, Arm B, Cohort 0 | Arm D | Dose Finding Phase, Arm C, Cohort 0 | Dose Finding Phase, Arm C, Cohort 1 | Dose Finding Phase, Arm D, Cohort 0 | Dose Finding Phase, Arm D, Cohort 1 | Dose Finding Phase, Arm D, Cohort 2 | Total
Number analyzed (Participants) | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7 | 52
Age, Continuous [Median (Full Range); unit: years] | 61 [52 to 69] | 48 [30 to 61] | 50 [37 to 68] | 52 [41 to 76] | 55 [48 to 83] | 62 [44 to 74] | 52 [49 to 70] | 57 [33 to 78] | 58 [27 to 65] | 55 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7 | 52
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 3 | 6 | 9 | 5 | 6 | 3 | 6 | 7 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  White | 4 | 3 | 4 | 5 | 5 | 6 | 2 | 6 | 5 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7 | 52

OUTCOME MEASURES:

1. Primary Outcome: Phase II Dose of BYL719/Alpelisib (Arm A and Arm B)
Description: Participants started BYL719 dose of 300mg daily for cohort 0. Consecutive cohorts were administered increasing or decreasing dose levels of BYL719. All participants within a cohort will be observed for toxicity for one cycle (28 days) prior to entering additional patients.
Time Frame: 28 days (1 Cycle)
Measure: Number; unit: mg
Groups:
- Arm A: BYL719 Plus Letrozole: For both the dose-finding phase and the expansion phase, patients may have stable or progressive disease on letrozole, and BYL719 will be added. A treatment cycle will consist of 28 days. Treatment doses for each AI will be fixed at the established dose. Patients will continue on treatment until progression of disease or unacceptable toxicity. The initial scan interval to assess disease status will be every two cycles (8 weeks) for the first four cycles (16 weeks), and then every 3rd cycle (12 weeks) thereafter.
  BYL719
  Letrozole
- Arm B: BYL719 Plus Exemestane: For both the dose-finding phase and the expansion phase, patients may have stable or progressive disease on Exemestane, and BYL719 will be added. A treatment cycle will consist of 28 days. Treatment doses for each AI will be fixed at the established dose. Patients will continue on treatment until progression of disease or unacceptable toxicity. The initial scan interval to assess disease status will be every two cycles (8 weeks) for the first four cycles (16 weeks), and then every 3rd cycle (12 weeks) thereafter.
  BYL719
  Exemestane
Arm/Group | Arm A: BYL719 Plus Letrozole | Arm B: BYL719 Plus Exemestane
Number analyzed (Participants) | 7 | 7
mg | 250 | 250

2. Primary Outcome: Phase II Dose of BYL719 (Arm C and Arm D)
Description: Participants started BYL719 dose of 250 daily for cohort 0. Consecutive cohorts were administered increasing or decreasing dose levels of BYL719.
Time Frame: 28 days (1 cycle)
Measure: Number; unit: mg
Groups:
- Arm C: BYL719 Plus Letrozole: For both the dose-finding and expansion phases of Arms C and D, patients may have stable or progressive disease on letrozole or exemestane, and BYL719 will be added.Letrozole 2.5mg orally once daily with BYL719 given on days 1-7 and 15-21 of a 28 day cycle. The starting dose of BYL719 in Arms C will be 250mg daily. Patients who are on study under Amendment 13, the scan interval will become every 4th cycle (16 weeks ±4 weeks) from their last scan.
  BYL719
  Letrozole
Arm/Group | Arm C: BYL719 Plus Letrozole | Arm D: BYL719 Plus Exemestane
Number analyzed (Participants) | 12 | 26
mg | 250 | 350

3. Secondary Outcome: Number of Participants Evaluated for Safety and Tolerability of BYL719 (Arm A, B, C and D)
Description: Toxicity will be tabulated using the NCI Common Toxicity Criteria (CTCAE), version 4.0. A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as at least possibly related to the study medication, meeting any of the criteria listed in the table below, and occurring during Cycle 1 (≤ 28 days following the first dose of BYL719, including those in which the event started in Cycle 1 and the confirmation of the DLT occurs in a subsequent cycle).
Time Frame: 28 days (1 cycle)
Measure: Count of Participants; unit: Participants
Groups:
- Arm C: BYL719 Plus Letrozole: DOSE FINDING PHASE, Arm B, Cohort 0: BYL719 300mg PO, Exemestane 25mg PO
Arm/Group | DOSE FINDING PHASE, Arm A, Cohort 0 | DOSE FINDING PHASE, Arm A, Cohort -1 | Arm C: BYL719 Plus Letrozole | Arm D | Dose Finding Phase, Arm C, Cohort 0 | Dose Finding Phase, Arm C, Cohort 1 | Dose Finding Phase, Arm D, Cohort 0 | Dose Finding Phase, Arm D, Cohort 1 | Dose Finding Phase, Arm D, Cohort 2
Number analyzed (Participants) | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7
Participants | 4 | 3 | 7 | 10 | 6 | 6 | 3 | 6 | 7

4. Secondary Outcome: Efficacy of BYL719 (Arm A, Arm B, Arm C and Arm D)
Description: Overall response rate
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: BYL719 Plus Letrozole | Arm B: BYL719 Plus Exemestane | Arm C: BYL719 Plus Letrozole | Arm D: BYL719 Plus Exemestane
Number analyzed (Participants) | 7 | 7 | 12 | 26
Participants
  Partial Response (PR) | 1 | 0 | 0 | 4
  Stable Disease (SD) | 4 | 3 | 6 | 13
  Progression of Disease (POD) | 0 | 3 | 1 | 5
  Complete Response (CR) | 0 | 0 | 0 | 1
  Unevaluable | 2 | 1 | 5 | 3

5. Secondary Outcome: Median Time to Treatment Failure/TTF
Description: Time to Treatment Failure/TTF defined as the time from on-study date to off-study date for any reason
Time Frame: through study completion, an average of 3.5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm A: BYL719 Plus Letrozole | Arm B: BYL719 Plus Exemestane | Arm C: BYL719 Plus Letrozole | Arm D: BYL719 Plus Exemestane
Number analyzed (Participants) | 7 | 7 | 12 | 26
weeks | 21 [2 to 169] | 8 [2 to 29] | 12 [3 to 72] | 17 [3 to 150]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | DOSE FINDING PHASE, Arm A, Cohort 0 | DOSE FINDING PHASE, Arm A, Cohort -1 | DOSE FINDING PHASE, Arm B, Cohort 0 | Arm D | Dose Finding Phase, Arm C, Cohort 0 | Dose Finding Phase, Arm C, Cohort 1 | Dose Finding Phase, Arm D, Cohort 0 | Dose Finding Phase, Arm D, Cohort 1 | Dose Finding Phase, Arm D, Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 2/7 | 0/10 | 1/6 | 0/6 | 0/3 | 0/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 4/7 | 2/10 | 3/6 | 2/6 | 0/3 | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 4/4 | 1/3 | 7/7 | 10/10 | 6/6 | 6/6 | 0/3 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DOSE FINDING PHASE, Arm A, Cohort 0 (N=4) | DOSE FINDING PHASE, Arm A, Cohort -1 (N=3) | DOSE FINDING PHASE, Arm B, Cohort 0 (N=7) | Arm D (N=10) | Dose Finding Phase, Arm C, Cohort 0 (N=6) | Dose Finding Phase, Arm C, Cohort 1 (N=6) | Dose Finding Phase, Arm D, Cohort 0 (N=3) | Dose Finding Phase, Arm D, Cohort 1 (N=6) | Dose Finding Phase, Arm D, Cohort 2 (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DOSE FINDING PHASE, Arm A, Cohort 0 (N=4) | DOSE FINDING PHASE, Arm A, Cohort -1 (N=3) | DOSE FINDING PHASE, Arm B, Cohort 0 (N=7) | Arm D (N=10) | Dose Finding Phase, Arm C, Cohort 0 (N=6) | Dose Finding Phase, Arm C, Cohort 1 (N=6) | Dose Finding Phase, Arm D, Cohort 0 (N=3) | Dose Finding Phase, Arm D, Cohort 1 (N=6) | Dose Finding Phase, Arm D, Cohort 2 (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2 | 2 | 2 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT01870505/Prot_SAP_000.pdf